CLINICAL TRIAL: NCT05281601
Title: Open-Label, Uncontrolled, Single Dose Study to Evaluate the Pharmacokinetics, Pharmacodynamics, and Safety of AZD7442 in Pediatric Participants Aged ≥ 29 Weeks Gestational Age to < 18 Years
Brief Title: AZD7442 Pharmacokinetics, Pharmacodynamics, and Safety Evaluation in Pediatrics
Acronym: TRUST
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D8850C00006; 2021-006056-13 (EudraCT Number)
Record Dates: First submitted 2022-02-16; First posted 2022-03-16 (Actual); Results first posted 2025-04-18 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: SARS-CoV-2
Keywords: AZD7442; Monoclonal antibodies (mAb); COVID-19; EVUSHELD
MeSH Terms: conditions — COVID-19 | interventions — cilgavimab and tixagevimab drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- AZD7442 (Experimental): All participants will receive a single dose of AZD7442 on Day 1, either IM (AZD8895 followed by AZD1061) or IV (AZD8895 + AZD1061 concurrently).
  Interventions: Drug: AZD7442

INTERVENTIONS:
Drug: AZD7442 — IM Administration: AZD8895 and AZD1061 (comprising AZD7442), must both be administered separately to the participant in a sequential order.
  IV Administration: AZD7442 is dosed by co-administration of AZD8895 and AZD1061 in a single IV infusion.
  Other Names: Evusheld

SUMMARY:
This study will evaluate the pharmacokinetics (PK), pharmacodynamics (PD), safety, and tolerability of AZD7442 administered intramuscularly (IM) or intravenously (IV) in pediatric participants aged ≥ 29 weeks GA to < 18 years.

DETAILED DESCRIPTION:
This is a Phase I, open-label, uncontrolled, multi-country, multi-center, single-dose study. Initially, 2 cohorts of participants will be enrolled: 1) participants who are severe acute respiratory syndrome coronavirus-2 (SARS-CoV-2) negative at screening and have not knowingly been exposed to a SARS-CoV-2 positive individual (pre-exposure prophylaxis); and 2) participants who are SARS-CoV-2 RT-PCR positive at screening and have mild to moderate COVID-19 symptoms. A third cohort might be added for the treatment of severe COVID-19. If included, this third cohort will include participants who are SARS-CoV-2 positive at screening and have severe COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be aged ≥ 29 weeks gestational age (GA) to < 18 years of age.
* Participant must weigh a minimum of 1.5 kg.

COHORT 1

* Increased risk of severe COVID-19 because of immunocompromised state or one or more comorbid conditions that increase the risk of severe COVID-19.
* Increased risk for SARS-CoV-2 infection.
* Medically stable (disease not requiring significant change in therapy or hospitalization for worsening disease during the one month prior to enrollment).
* A negative RT-PCR test collected ≤ 3 days prior to Day 1 or a negative rapid SARS-CoV-2 antigen test at screening.
* No COVID-19 symptoms prior to enrollment within 10 days of dosing.
* Increased risk for SARS-CoV-2 infection.

COHORT 2

* Increased risk of severe COVID-19 because of immunocompromised state or one or more comorbid conditions that increase the risk of severe COVID-19.
* Medically stable (disease not requiring significant change in therapy or hospitalization for worsening disease during the one month prior to enrollment).
* A positive RT-PCR test collected ≤ 3 days prior to Day 1 or a positive rapid SARS-CoV-2 antigen test at screening.
* Symptomatic participants must be dosed with IMP no more than 7 days from the self-reported date of first reported sign/symptom.
* Oxygenation saturation of ≥ 92% obtained at rest within 24 hours prior to Day 1 unless the potential participant regularly receives chronic supplementary oxygen for an underlying lung condition.

Note that Cohort 2 will only be included if the indication is progressed in adults.

COHORT 3

* Participants hospitalized with COVID-19 with a time between onset of symptoms and dosing AZD7442 of ≤ 7 days.
* A positive RT-PCR test collected ≤ 3 days before Day 1 or a positive rapid SARS-CoV-2 antigen test at screening.
* Spontaneous blood Alanine Aminotransferase (ALT)/Aspartate Transaminase (AST) levels ≤ 5 times the ULN.
* Glomerular Filtration Rate (GFR) ≥ 30 mL/min/1.73 m2.

Participants will receive IM AZD7442 unless they meet any of the following criteria for IV administration:

* The participant has severe COVID-19.
* Contraindication of intramuscular (IM) dose due to thrombocytopenia, coagulation defects or any other condition that would compromise the absorption of AZD7442 or safety of the participant.
* Physician considers IV the appropriate route.

Exclusion Criteria:

All Cohorts

* Cohort 1: Significant infection or other acute illnesses including fever on or the day prior to receiving AZD7442.
* History of SARS-CoV-1 or Middle East Respiratory Syndrome Coronavirus (MERS-CoV).
* Cohorts 1 and 2: Current need for immediate medical attention or current need for hospitalization.
* Mechanical ventilation or extracorporeal membrane oxygenation requirement for COVID-19.
* History of allergic or reaction to any component of the study drug formulation.
* History of hypersensitivity, injection/infusion-relation reactions or severe adverse reactions following administration of a monoclonal antibody (mAb).
* Co-morbidity requiring surgery within 7 days prior to study entry or is deemed life-threatening within 30 days prior to study entry.
* Prior receipt of convalescent COVID-19 plasma/sera or hyperimmune globulin therapy.
* Prior receipt of mAb/biologic indicated for the prevention of SARS-CoV-2, treatment of COVID-19, or expected receipt during the period of study follow-up.
* Prior receipt of a COVID-19 vaccine ≤ 14 days before screening or plan to receive a COVID-19 vaccination ≤ 14 days after IMP administration at study Visit 1.
* History of alcohol or drug abuse within the past 2 years.
* Investigational Drugs or Devices: Treatment with investigational drug or device in another clinical trial within the last 30 days or 5 half-lives of the drug (whichever is longer) prior to screening. Note: Participation in observational studies (ie, studies that do not require medication, blood draws, or an additional intervention) is not exclusionary. Interventional trials which do not include investigational drugs (only include approved therapies), or investigational treatment regimens may be considered if the blood draw requirements and study interventions are minimal and not deemed by the Investigator to interfere with completion of the planned study sampling and follow-up.
* Vulnerable persons (eg, ward of the state, kept in detention).

Ages: 0 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 46 (Actual)
Dates: Start 2022-03-21 (Actual); Primary Completion 2024-04-16 (Actual); Study Completion 2024-04-16 (Actual)

CONTACTS AND LOCATIONS:
Locations (11):
- United States (7):
  - Research Site, Long Beach, California
  - Research Site, Aurora, Colorado
  - Research Site, Washington D.C., District of Columbia
  - Research Site, Idaho Falls, Idaho
  - Research Site, Stony Brook, New York
  - Research Site, Providence, Rhode Island
  - Research Site, Mt. Pleasant, South Carolina
- Research Site, Leuven, Belgium
- Research Site, Belo Horizonte, Brazil
- Research Site, Frankfurt am Main, Germany
- Research Site, Southampton, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: D8850C00006_Redacted_CSP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D8850C00006&attachmentIdentifier=d2a6d8c2-f8a7-4c36-b807-1571ec897378&fileName=D8850C00006_Redacted_CSP.pdf&versionIdentifier=
- See also: D8850C00006_Redacted_CSR_Synopsi — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D8850C00006&attachmentIdentifier=88d5eb25-82fe-442e-ad6f-fa3495442908&fileName=D8850C00006_Redacted_CSR_Synopsis.pdf&versionIdentifier=
- See also: D8850C00006_Redacted_SAP. — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D8850C00006&attachmentIdentifier=a58e68e3-e288-4a23-8e31-1765c89975f5&fileName=D8850C00006_Redacted_SAP.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted from 21 March 2022 to 16 April 2024 at 11 sites in 5 countries worldwide.
Pre-assignment Details: Participants who met the inclusion criteria and none of the exclusion criteria were enrolled to the study. All study assessments were performed as per the schedule of assessment.
Groups:
- Cohort 1: Participants who were SARS-CoV-2 RT-PCR negative received single dose of AZD7442 on Day 1, either as intramuscularly (IM) (AZD8895 followed by AZD1061) or as intravenously (IV) (AZD8895 + AZD1061 concurrently)
- Cohort 2: Participants who were SARS-CoV-2 RT-PCR positive received single dose of AZD7442 on Day 1, either as IM (AZD8895 followed by AZD1061) or as IV (AZD8895 + AZD1061 concurrently).
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2
Started | 44 | 2
Completed | 37 | 1
Not Completed | 7 | 1
Not completed — Physician Decision | 2 | 0
Not completed — Lost to Follow-up | 2 | 0
Not completed — Death | 1 | 0
Not completed — Withdrawal by parent/guardian | 2 | 1

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set (SAF) consisted of all participants who had received investigational medicinal product (IMP).
Groups:
- Cohort 1: Participants who were SARS-CoV-2 RT-PCR negative received single dose of AZD7442 on Day 1, either as IM (AZD8895 followed by AZD1061) or as IV (AZD8895 + AZD1061 concurrently)
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Total
Number analyzed (Participants) | 44 | 2 | 46
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 44 | 2 | 46
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 0 | 25
  Male | 19 | 2 | 21
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Black or African American | 11 | 0 | 11
  Race: Multiple | 2 | 0 | 2
  Race: Not Reported | 2 | 1 | 3
  Race: White | 28 | 0 | 28
  Race: Other | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Serum Concentrations of AZD7442
Description: The serum concentrations of AZD7442 after a single IM or IV dose in pediatric participants were evaluated. The serum concentrations for each scheduled time point were summarized by route of administration using appropriate descriptive statistics, based on the (Pharmacokinetic analysis) PK analysis set.
Time Frame: IM - Day 4, Day 8, Day 11, Day 15 and Day 366; IV - Day 1, Day 4, Day 8, Day 11, Day 15 and Day 366
Population: The PK set consisted of all participants who received AZD7442 and from whom PK blood samples were assumed not to be affected by factors such as protocol violations, and who had at least one quantifiable serum PK observation post-dose.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram per milliliter (ug/mL)
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 20 | 1
Microgram per milliliter (ug/mL)
  Day 4 AZD7442 intramuscular: number analyzed (Participants) | 8 | 0
  Day 4 AZD7442 intramuscular | 86.32 (72.72) |
  Day 8 AZD7442 intramuscular: number analyzed (Participants) | 4 | 0
  Day 8 AZD7442 intramuscular | 91.88 (86.03) |
  Day 11 AZD7442 intramuscular: number analyzed (Participants) | 5 | 0
  Day 11 AZD7442 intramuscular | 92.49 (20.91) |
  Day 15 AZD7442 intramuscular: number analyzed (Participants) | 7 | 0
  Day 15 AZD7442 intramuscular | 84.69 (33.69) |
  Day 366 AZD7442 intramuscular: number analyzed (Participants) | 20 | 0
  Day 366 AZD7442 intramuscular | 4.084 (57.91) |
  Day 1 AZD7442 intravenous: number analyzed (Participants) | 17 | 1
  Day 1 AZD7442 intravenous | 199.9 (23.16) | NA (NA) — Data were not reported due to presence of insufficient number of participants at that timepoint for analysis as is pre-specified in SAP.
  Day 4 AZD7442 intravenous: number analyzed (Participants) | 3 | 0
  Day 4 AZD7442 intravenous | NA (NA) — Data were not reported due to presence of insufficient number of participants at that timepoint for analysis as is pre-specified in SAP. |
  Day 8 AZD7442 intravenous: number analyzed (Participants) | 6 | 0
  Day 8 AZD7442 intravenous | 89.47 (30.60) |
  Day 11 AZD7442 intravenous: number analyzed (Participants) | 6 | 0
  Day 11 AZD7442 intravenous | 95.02 (20.35) |
  Day 15 AZD7442 intravenous: number analyzed (Participants) | 3 | 1
  Day 15 AZD7442 intravenous | NA (NA) — Data were not reported due to presence of insufficient number of participants at that timepoint for analysis as is pre-specified in SAP. | NA (NA) — Data were not reported due to presence of insufficient number of participants at that timepoint for analysis as is pre-specified in SAP.
  Day 366 AZD7442 intravenous: number analyzed (Participants) | 13 | 1
  Day 366 AZD7442 intravenous | 2.047 (74.56) | NA (NA) — Data were not reported due to presence of insufficient number of participants at that timepoint for analysis as is pre-specified in SAP.

2. Primary Outcome: Maximum Serum Concentration (Cmax)
Description: The Cmax of AZD7442 after a single IM or IV dose in pediatric participants was evaluated. The PK parameters were summarized by route of administration using appropriate descriptive statistics based on the PK analysis set.
Time Frame: Day 1 to Day 366 or early discontinuation visit (approximately [approx.] 24 months)
Population: The PK analysis set consisted of all participants who received AZD7442 and from whom PK blood samples were assumed not to be affected by factors such as protocol violations, and who had at least one quantifiable serum PK observation post-dose.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram per milliliter (ug/mL)
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 24 | 1
Microgram per milliliter (ug/mL)
  AZD7442 intramuscular: number analyzed (Participants) | 24 | 0
  AZD7442 intramuscular | 92.47 (44.22) |
  AZD7442 intravenous: number analyzed (Participants) | 19 | 1
  AZD7442 intravenous | 189.3 (27.72) | NA (NA) — Data were not reported due to presence of insufficient number of participants at that timepoint for analysis as is pre-specified in SAP.

3. Primary Outcome: Time to Reach Maximum Serum Concentration (Tmax)
Description: The tmax of AZD7442 after a single IM or IV dose in pediatric participants was evaluated. The PK parameters were summarized by route of administration using appropriate descriptive statistics based on the PK analysis set.
Time Frame: Day 1 to Day 366 or early discontinuation visit (approx. 24 months)
Population: as for outcome 2
Measure: Median (Full Range); unit: Day
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 24 | 1
Day
  AZD7442 intramuscular: number analyzed (Participants) | 24 | 0
  AZD7442 intramuscular | 11.44 [0.76 to 32.73] |
  AZD7442 intravenous: number analyzed (Participants) | 19 | 1
  AZD7442 intravenous | 0.01 [0.01 to 9.95] | NA [0.01 to 0.01] — Data were not reported due to presence of insufficient number of participants at that timepoint for analysis as is pre-specified in SAP.

4. Primary Outcome: Terminal Half-life (t1/2)
Description: The t1/2 of AZD7442 after a single IM or IV dose in pediatric participants was evaluated. The PK parameters were summarized by route of administration using appropriate descriptive statistics based on the PK analysis set.
Time Frame: Day 1 to Day 366 or early discontinuation visit (approx. 24 months)
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Day
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 22 | 1
Day
  AZD7442 intramuscular: number analyzed (Participants) | 22 | 0
  AZD7442 intramuscular | 78.95 (24.21) |
  AZD7442 intravenous: number analyzed (Participants) | 17 | 1
  AZD7442 intravenous | 65.61 (22.38) | NA (NA) — Data were not reported due to presence of insufficient number of participants at that timepoint for analysis as is pre-specified in SAP.

5. Primary Outcome: Area Under the Serum Concentration Versus Time Curve From Time Zero to Time of Last Measurable Concentration (AUC0-last)
Description: The AUC0-last of AZD7442 after a single IM or IV dose in pediatric participants was evaluated. The PK parameters were summarized by route of administration using appropriate descriptive statistics based on the PK analysis set.
Time Frame: Day 1 to Day 366 or early discontinuation visit (approx. 24 months)
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Day*ug/mL
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 23 | 1
Day*ug/mL
  AZD7442 intramuscular: number analyzed (Participants) | 23 | 0
  AZD7442 intramuscular | 9884 (42.84) |
  AZD7442 intravenous: number analyzed (Participants) | 19 | 1
  AZD7442 intravenous | 9342 (36.45) | NA (NA) — Data were not reported due to presence of insufficient number of participants at that timepoint for analysis as is pre-specified in SAP.

6. Primary Outcome: Area Under the Serum Concentration Versus Time Curve Extrapolated to Infinity (AUC0-inf)
Description: The AUC0-inf of AZD7442 after a single IM or IV dose in pediatric participants was evaluated. The PK parameters were summarized by route of administration using appropriate descriptive statistics based on the PK analysis set.
Time Frame: Day 1 to Day 366 or early discontinuation visit (approx. 24 months)
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Day*ug/mL
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 22 | 1
Day*ug/mL
  AZD7442 intramuscular: number analyzed (Participants) | 22 | 0
  AZD7442 intramuscular | 11000 (38.03) |
  AZD7442 intravenous: number analyzed (Participants) | 17 | 1
  AZD7442 intravenous | 10870 (21.09) | NA (NA) — Data were not reported due to presence of insufficient number of participants at that timepoint for analysis as is pre-specified in SAP.

7. Primary Outcome: Time to Last Measurable Concentration (Tlast)
Description: The tlast of AZD7442 after a single IM or IV dose in pediatric participants was evaluated. The PK parameters were summarized by route of administration using appropriate descriptive statistics based on the PK analysis set.
Time Frame: Day 1 to Day 366 or early discontinuation visit (approx. 24 months)
Population: as for outcome 2
Measure: Median (Full Range); unit: Day
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 24 | 1
Day
  AZD7442 intramuscular: number analyzed (Participants) | 24 | 0
  AZD7442 intramuscular | 351.38 [0.76 to 401.00] |
  AZD7442 intravenous: number analyzed (Participants) | 19 | 1
  AZD7442 intravenous | 355.97 [33.81 to 377.26] | NA [354.90 to 354.90] — Data were not reported due to presence of insufficient number of participants at that timepoint for analysis as is pre-specified in SAP.

8. Primary Outcome: Percentage of AUC0-inf Extrapolated to Infinity (% AUCex)
Description: The %AUCex of AZD7442 after a single IM or IV dose in pediatric participants was evaluated. The PK parameters were summarized by route of administration using appropriate descriptive statistics based on the PK analysis set.
Time Frame: Day 1 to Day 366 or early discontinuation visit (approx. 24 months)
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percentage of AUC extrapolated to ∞
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 22 | 1
Percentage of AUC extrapolated to ∞
  AZD7442 intramuscular: number analyzed (Participants) | 22 | 0
  AZD7442 intramuscular | 4.799 (78.26) |
  AZD7442 intravenous: number analyzed (Participants) | 17 | 1
  AZD7442 intravenous | 3.018 (179.9) | NA (NA) — Data were not reported due to presence of insufficient number of participants at that timepoint for analysis as is pre-specified in SAP.

9. Primary Outcome: Apparent Total Clearance (CL/F)
Description: The CL/F of AZD7442 after a single IM dose in pediatric participants was evaluated. The PK parameters were summarized by route of administration using appropriate descriptive statistics based on the PK analysis set.
Time Frame: Day 1 to Day 366 or early discontinuation visit (approx. 24 months)
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter/day
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 22 | 0
Liter/day | 0.04807 (75.26) |

10. Primary Outcome: Apparent Volume of Distribution Based on Terminal Phase (Vz/F)
Description: The Vz/F of AZD7442 after a single IM dose in pediatric participants was evaluated. The PK parameters were summarized by route of administration using appropriate descriptive statistics based on the PK analysis set.
Time Frame: Day 1 to Day 366 or early discontinuation visit (approx. 24 months)
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 22 | 0
Liter | 5.475 (98.74) |

11. Primary Outcome: Systemic Clearance (CL)
Description: The CL of AZD7442 after a single IV dose in pediatric participants was evaluated. The PK parameters were summarized by route of administration using appropriate descriptive statistics based on the PK analysis set.
Time Frame: Day 1 to Day 366 or early discontinuation visit (approx. 24 months)
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter/day
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 17 | 1
Liter/day | 0.02759 (21.09) | NA (NA) — Data were not reported due to presence of insufficient number of participants at that timepoint for analysis as is pre-specified in SAP.

12. Primary Outcome: Volume of Distribution at Steady State (Vss)
Description: The Vss of AZD7442 after a single IV dose in pediatric participants was evaluated. The PK parameters were summarized by route of administration using appropriate descriptive statistics based on the PK analysis set.
Time Frame: Day 1 to Day 366 or early discontinuation visit (approx. 24 months)
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 17 | 1
Liter | 2.605 (20.34) | NA (NA) — Data were not reported due to presence of insufficient number of participants at that timepoint for analysis as is pre-specified in SAP.

13. Primary Outcome: Number of Participants With Adverse Events (AE)
Description: The safety and tolerability of AZD7442 after a single IM or IV dose in pediatric participants was evaluated.
Time Frame: Day 1 to Day 366 or early discontinuation visit (approx. 24 months)
Population: The SAF consisted of all participants who had received IMP.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 44 | 2
Participants
  Any AE | 39 | 2
  Any Serious Adverse Event (SAE) | 8 | 1
  Any Severe AE | 6 | 0
  Any SAE with outcome death | 1 | 0
  Any AE leading to study discontinuation | 0 | 0
  Any possibly related AE | 3 | 0
  Any possibly related SAE | 0 | 0
  Any possibly related Severe AE | 0 | 0
  Any possibly related Adverse Event of Special interest (AESI) | 1 | 0

14. Secondary Outcome: Number of Participants With Positive Antidrug Antibodies (ADA) Result to AZD7442.
Description: The immunogenicity profile of AZD7442 after a single IM or IV dose in pediatric participants was evaluated.
  A participant is defined as ADA-positive to AZD7442 if they have a positive ADA result to AZD8895 and/or AZD1061 at any time, including baseline and all postbaseline.
Time Frame: Day 1 to Day 366 or early discontinuation visit (approx. 24 months)
Population: The AZD7442 ADA Evaluable Analysis Set (ADS3) consisted of all participants who were AZD8895 ADA evaluable and/or AZD1061 ADA evaluable.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 44 | 2
Participants
  AZD7442 intramuscular ADA positive subject | 2 | 0
  AZD7442 intravenous ADA positive subject | 2 | 0

15. Primary Outcome: Number of Participants With Adverse Event of Special Interest (AESI)
Description: Number of pediatric participants with AESI after a single IM or IV dose were evaluated.
  An AESI is a pre-specified medically significant event that has the potential to be causally associated with a vaccine product.
Time Frame: Day 1 to day 366 or early discontinuation visit (approx. 24 months)
Population: The SAF consisted of all participants who had received IMP.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 44 | 2
Participants | 1 [0.1 to 12.0] | 0 [0 to 0]

16. Secondary Outcome: Cohort 2 - Percentage of Participants With Progression of COVID-19 Through Day 29
Description: Percentage of participants with progression of COVID-19 through Day 29 in Cohort 2 in pediatric participants was evaluated.
Time Frame: Day 1 to Day 366 or early discontinuation visit (approx. 24 months)
Population: The SAF consisted of all participants who had received IMP.
Measure: Number; unit: Percentage of participants
Arm/Group | Cohort 2
Number analyzed (Participants) | 2
Percentage of participants | 0

17. Secondary Outcome: Cohort 2 - Number of Participants With COVID-19 Related Death Occurring After Dosing With IMP Through 90 Days
Description: Number of participants with COVID-19 related death occurring after dosing with IMP through 90 days in Cohort 2 in pediatric participants were evaluated.
Time Frame: Day 1 to Day 366 or early discontinuation visit (approx. 24 months)
Population: The SAF consisted of all participants who had received IMP.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 2
Number analyzed (Participants) | 2
Participants | 0

18. Secondary Outcome: Titre of SARS-CoV-2 Neutralizing Antibodies
Description: The pharmacodynamics of AZD7442 after a single dose in pediatric participants was evaluated.
  The result for overall vaccination status were presented.
Time Frame: Day 31 to Day 366 or early discontinuation visit (approx. 24 months)
Population: The SARS-CoV-2 nAb Evaluable Analysis Set (SES) consisted of all participants in the Safety Analysis Set from whom blood samples were assumed not to be affected by factors such as protocol violations, and who had at least one quantifiable serum titer observation post dose.
Measure: Geometric Mean (Full Range); unit: ug/mL
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 23 | 1
ug/mL
  Intramuscular Day 31: number analyzed (Participants) | 23 | 0
  Intramuscular Day 31 | 52720 [355 to 139000] |
  Intramuscular Day 366: number analyzed (Participants) | 22 | 0
  Intramuscular Day 366 | 1699 [143 to 4340] |
  Intravenous Day 31: number analyzed (Participants) | 18 | 1
  Intravenous Day 31 | 52950 [20800 to 120000] | NA [19800 to 19800] — Data were not reported due to presence of insufficient number of participants at that timepoint for analysis as is pre-specified in SAP.
  Intravenous Day 366: number analyzed (Participants) | 11 | 1
  Intravenous Day 366 | 1078 [398 to 4460] | NA [252 to 252] — Data were not reported due to presence of insufficient number of participants at that timepoint for analysis as is pre-specified in SAP.

19. Secondary Outcome: Cohort 1 (Prophylaxis) - Number of Participants With SARS-CoV-2 Infections
Description: Number of participants with SARS-CoV-2 infections with or without COVID-19 symptoms after a single IM or IV dose of AZD7442 in pediatric participants were evaluated.
Time Frame: Day 1 to Day 366 or early discontinuation visit (approx. 24 months)
Population: The SAF consisted of all participants who had received IMP.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1
Number analyzed (Participants) | 44
Participants
  Overall | 10
  Intramuscular administration | 7
  Intravenous administration | 3

ADVERSE EVENTS:
Time Frame: Day 1 to Day 366 or early discontinuation visit (approx. 24 months)
Description: The SAF consisted of all participants who had received IMP.
Arm/Group | Cohort 1 | Cohort 2
All-Cause Mortality (participants affected / at risk) | 1/44 | 0/2
Serious Adverse Events (participants affected / at risk) | 8/44 | 1/2
Other Adverse Events (participants affected / at risk) | 34/44 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=44) | Cohort 2 (N=2)
Croup infectious (Infections and infestations) | 1 (1) | 0 (0)
Device related sepsis (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis Escherichia coli (Infections and infestations) | 1 (1) | 0 (0)
Lower respiratory tract infection bacterial (Infections and infestations) | 1 (1) | 0 (0)
Metapneumovirus infection (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection viral (Infections and infestations) | 1 (1) | 0 (0)
Rhinovirus infection (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Febrile bone marrow aplasia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (5) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 1 (1) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Epilepsy (Nervous system disorders) | 0 (0) | 1 (1)
Nephrotic syndrome (Renal and urinary disorders) | 1 (1) | 0 (0)
Ovarian cyst ruptured (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Henoch-Schonlein purpura (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=44) | Cohort 2 (N=2)
Upper respiratory tract infection (Infections and infestations) | 12 (27) | 0 (0)
Viral infection (Infections and infestations) | 11 (13) | 0 (0)
COVID-19 (Infections and infestations) | 10 (10) | 0 (0)
Acute sinusitis (Infections and infestations) | 4 (7) | 0 (0)
Otitis media acute (Infections and infestations) | 4 (4) | 0 (0)
Pharyngitis streptococcal (Infections and infestations) | 4 (4) | 0 (0)
Influenza (Infections and infestations) | 3 (3) | 0 (0)
Nasopharyngitis (Infections and infestations) | 3 (7) | 0 (0)
Ear infection (Infections and infestations) | 0 (0) | 1 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 0 (0)
Nausea (Gastrointestinal disorders) | 4 (4) | 0 (0)
Vomiting (Gastrointestinal disorders) | 4 (4) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 0 (0)
Headache (Nervous system disorders) | 4 (4) | 0 (0)
SARS-CoV-2 test positive (Investigations) | 3 (3) | 0 (0)
Influenza A virus test positive (Investigations) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 7 (13) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No unpublished information may be disclosed without prior written approval from AstraZeneca.

DOCUMENTS (2):
  • Study Protocol (2023-10-25): https://cdn.clinicaltrials.gov/large-docs/01/NCT05281601/Prot_000.pdf
  • Statistical Analysis Plan (2023-07-31): https://cdn.clinicaltrials.gov/large-docs/01/NCT05281601/SAP_001.pdf